CLINICAL TRIAL: NCT03062033
Title: Real-World Evaluation Screening Study and Registry of Dyskinesia in Patients Taking Antipsychotic Agents
Acronym: RE-Kinect
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Evidera (Industry)
Responsible Party: Sponsor
Other Study IDs: EVA-19350
Record Dates: First submitted 2017-02-03; First posted 2017-02-23 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Patients without visible signs of involuntary movements (possible TD) at time of clinician assessment
- Cohort 2: Patients with visible signs of involuntary movements (possible TD) at the time of clinician assessment

SUMMARY:
Prospective study to quantify the prevalence of possible tardive dyskinesia (TD) in outpatient psychiatry practices in the United States (US), as well as to describe the associated disease burden in a cohort of patients with one or more psychiatric disorders and a cumulative lifetime exposure to antipsychotic medication of three months or more.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a cumulative lifetime exposure to antipsychotic medication of three months or more
* Patient has a clinician confirmed diagnosis of one or more psychiatric disorder(s), as defined in the DSM-5
* Patient has a usual care clinic visit scheduled during the study recruitment window (i.e. a pre-defined 2-week period)
* Patient is able to read and understand English
* Patient is willing and able to comply with the study requirements

Exclusion Criteria:

* Patient is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be 18 years or older with a cumulative lifetime exposure to antipsychotic medication of three months or more.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Customized clinician-reported outcomes | 12 months
  Clinician evaluation of patient burden due to tardive dyskinesia symptoms
EuroQOL 5 Dimensions EQ-5D-5L) | 12 months
  General, single index measure for describing and valuing health-related quality of life.
Customized caregiver-reported outcomes: | 12 months
  Caregiver evaluation of perceived burden of symptoms on patients as well as the impact on the caregiver
Sheehan Disability Scale (SDS) | 12 months
  Assessment of functional impairment and disability

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — Chief Medical Officer
Locations (32):
- United States (32):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Long Beach, California
  - Neurocrine Clinical Site, Los Gatos, California
  - Neurocrine Clinical Site, Oceanside, California
  - Neurocrine Clinical Site, Gainesville, Florida
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Jacksonville, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Miami Beach, Florida
  - Neurocrine Clinical Site, Miami Springs, Florida
  - Neurocrine Clinical Site, North Miami, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Decatur, Georgia
  - Neurocrine Clinical Site, Honolulu, Hawaii
  - Neurocrine Clinical Site, Naperville, Illinois
  - Neurocrine Clinical Site, Michigan City, Indiana
  - Neurocrine Clinical Site, Grand Rapids, Michigan
  - Neurocrine Clinical Site, Rochester, Michigan
  - Neurocrine Clinical Site, Kansas City, Missouri
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Nashua, New Hampshire
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Hickory, North Carolina
  - Neurocrine Clinical Site, Garfield Heights, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, San Antonio, Texas
  - Neurocrine Clinical Site, Salt Lake City, Utah
  - Neurocrine Clinical Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No